CLINICAL TRIAL: NCT03688906
Title: Specimen Collection Study for Cancer
Brief Title: AI-EMERGE: Development and Validation of a Multi-analyte, Blood-based Colorectal Cancer Screening Test
Status: Completed | Type: Observational
Sponsor: Freenome Holdings Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AI-EMERGE/FRE-001
Record Dates: First submitted 2018-08-27; First posted 2018-09-28 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Colo-rectal Cancer; Cancer Colon; Cancer, Rectum; Neoplasms,Colorectal; Polyps; Polyp of Colon; Adenoma; Adenoma Colon
Keywords: Liquid biopsy; Blood test cancer; Cancer diagnostic; Genomics; Genomic test; AI genomics; CRC; Cancer screening
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms; Polyps; Colonic Polyps; Adenoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort A: Blood and stool specimen collection.
  Study samples must be collected prior to any treatment.
- Cohort B: Blood and stool specimen collection.
  Samples must be collected prior to performing bowel preparation for the colonoscopy.
- Cohort C: Blood and stool specimen collection.
  Study samples must be collected prior to any treatment.

SUMMARY:
Freenome is using a type of artificial intelligence, called machine learning, to identify patterns of cell-free biomarkers in blood to detect cancer early. The purpose of this study is to develop and validate a blood-based assay to detect colorectal cancer by collecting blood and stool samples from healthy patients undergoing routine screening colonoscopy and from patients recently diagnosed with colorectal cancer or advanced adenomas.

DETAILED DESCRIPTION:
Early detection of cancer combined with effective treatment improves survival and quality of life. Freenome is using a type of artificial intelligence, called machine learning, to identify patterns of cell-free biomarkers in the blood to detect cancer early. The purpose of this study is to develop and validate a blood-based assay for the early detection of colorectal cancer. The study will collect blood and stool samples from healthy patients undergoing routine screening colonoscopy and from patients recently diagnosed with colorectal cancer or advanced adenomas. A blood-based test for colorectal cancer and pre-cancerous lesions could offer an accurate, convenient, and patient-friendly screening option for current and future generations, and, in doing so, could save and improve lives by increasing adherence and early detection.

Freenome is looking for three types of patients in this study:

Cohort A:

People ages 50-84 who have been recently diagnosed with (or strong clinical suspicion for) colorectal cancer or advanced adenoma. Blood samples must be collected before any cancer treatment has been initiated.

Cohort B:

People ages 50-84 undergoing routine screening colonoscopies for colorectal cancer as part of their regular medical check-ups. Blood samples must be collected before bowel preparation for the colonoscopy.

Cohort C:

People 18 years or older who have been recently diagnosed with (or strong clinical suspicion for) colorectal cancer or advanced adenoma. Blood samples must be collected before any cancer treatment has been initiated.

ELIGIBILITY:
COHORT A

Inclusion Criteria:

* 50-84 years of age (inclusive) at the time of screening
* Recently diagnosed with (or strong clinical suspicion for) primary colorectal cancer or advanced adenoma with plans to surgically or endoscopically remove the target lesion(s)
* At least 7 days before but no more than 6 months after the most recent colonoscopy
* Able and willing to provide blood and stool (optional) samples per protocol
* Able to comprehend and willing to sign and date the written informed consent document(s) and any applicable medical record release documents for the study

Key Exclusion Criteria:

* Personal history of colorectal cancer, colorectal adenomas (excluding non-adenomatous (e.g., hyperplastic polyps)) or aerodigestive tract cancer (other than most recent diagnosis)
* Colonoscopy within the previous 9 years (other than most recent diagnosis)
* Overt rectal bleeding within the previous 30 days
* Have a medical condition which, in the opinion of the investigator, should preclude enrollment into the study.
* Have participated or be currently participating in a clinical research study in which an experimental medication has been administered during the 60 days up to and including the date of providing informed consent or may be administered through the time of the colonoscopy.
* If female, known to be pregnant.

COHORT B

Inclusion Criteria:

* 50-84 years of age (inclusive) at the time of screening
* Planning to undergo a screening colonoscopy within 75 days after providing signed informed consent
* Able and willing to provide blood and stool (optional) samples per protocol
* Able to comprehend and willing to sign and date the written informed consent document(s) and any applicable medical record release documents for the study

Key Exclusion Criteria:

* Personal history of colorectal cancer, colorectal adenoma (excluding non-adenomatous (e.g., hyperplastic polyps)) or aerodigestive tract cancer
* Colonoscopy within the previous 9 years
* Overt rectal bleeding within the previous 30 days
* Have a medical condition which, in the opinion of the investigator, should preclude enrollment into the study.
* Have participated or be currently participating in a clinical research study in which an experimental medication has been administered during the 60 days up to and including the date of providing informed consent or may be administered through the time of the colonoscopy.
* If female, known to be pregnant.

COHORT C

Inclusion Criteria:

* At least 18 years of age (inclusive) at the time of screening
* Recently diagnosed with (or strong clinical suspicion for) primary colorectal cancer or advanced adenoma with plans to surgically or endoscopically remove the target lesion(s)
* At least 7 days before but no more than 6 months after the most recent colonoscopy
* Able and willing to provide blood and stool (optional) samples per protocol
* Able to comprehend and willing to sign and date the written informed consent document(s) and any applicable medical record release documents for the study

Exclusion Criteria:

* Have a medical condition which, in the opinion of the investigator, should preclude enrollment into the study.
* Have participated or be currently participating in a clinical research study in which an experimental medication has been administered during the 60 days up to and including the date of providing informed consent or may be administered through the time of the colonoscopy.
* If female, be known to be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects for the study will be enrolled into three cohorts:
  * Cohort (A): People ages 50-84 who have been recently diagnosed with (or strong clinical suspicion for) colorectal cancer or advanced adenoma. Blood samples must be collected before any cancer treatment has been initiated.
  * Cohort (B): People ages 50-84 undergoing routine screening colonoscopies for colorectal cancer as part of their regular medical check-ups. Blood samples must be collected before bowel preparation for the colonoscopy.
  * Cohort (C): People 18 years or older who have been recently diagnosed with (or strong clinical suspicion for) colorectal cancer or advanced adenoma. Blood samples must be collected before any cancer treatment has been initiated.
Sampling Method: Non-Probability Sample
Enrollment: 3275 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Diagnosis of colorectal cancer or advanced adenomas in patients undergoing routine screening colonoscopy, or post-colonoscopy | 6 months
  Clinically annotated plasma samples from participants will undergo multi-omic analyses to characterize cell-free biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Girish Putcha, M.D., Ph.D, Principal Investigator — Freenome Holdings Inc.
Locations (30):
- United States (29):
  - Clinical Research Associates, Huntsville, Alabama
  - Del Sol Research Management, Chandler, Arizona
  - Del Sol Research Management,, Tucson, Arizona
  - Del Sol Research Management, Tucson, Arizona
  - Preferred Research Partners, Little Rock, Arkansas
  - Precision Research Institute, Chula Vista, California
  - Diverse Research Solutions, Oxnard, California
  - Precision Research Institute, San Diego, California
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - Palmetto Research, Hialeah, Florida
  - Clinical Research of Homestead, Homestead, Florida
  - Advanced Gastroenterology Associates, LLC, Palm Harbor, Florida
  - Rockford Gastroenterology, Rockford, Illinois
  - Delta Research Partners, Bastrop, Louisiana
  - New Orleans Research Institute, Metairie, Louisiana
  - Louisiana Research Center, Shreveport, Louisiana
  - Commonwealth Clinical Studies, Brockton, Massachusetts
  - Quality Clinical Research, Omaha, Nebraska
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cumberland Research Associates, Fayetteville, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Trial Management Associates, Wilmington, North Carolina
  - The Jackson Clinic, Jackson, Tennessee
  - Advanced Research Institute, Ogden, Utah
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Verity Research Inc, Fairfax, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Washington Gastroenterology, Bellevue, Washington
- Forzani and MacPhail Colon Cancer Screening Centre, Calgary, Alberta, Canada

REFERENCES:
- [Result] Putcha G, Liu T-Y, Ariazi E, Bertin M, Drake A, Dzamba M, Hogan G, Kothen-Hill S, Liao J, Li K, Mahajan S, Palaniappan K, Sansanwal P, St John J, Ulz P, Wan N, Warsinske H, Weinberg D, Yang R, Lin J. Blood-based detection of early-stage colorectal cancer using multiomics and machine learning. [Abstract] J Clin Oncol 38 (Suppl 4): A-66, 2020.